CLINICAL TRIAL: NCT01430338
Title: Different Metabolic Characteristics in the Presence of Brown Adipose Tissue in Humans
Status: Completed | Type: Observational
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, K. M. Choi, Professor, Korea University
Other Study IDs: BAT
Record Dates: First submitted 2011-08-24; First posted 2011-09-08 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2011-09

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — plasma and serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- BAT: brown adipose tissue detected, undetected

SUMMARY:
Functional brown adipose tissue (BAT) exists in adult humans and can be detected by PET and especially during acute cold exposure. It is conceivable that BAT activity might reduce the risk of developing obesity since fat stores are used for thermogenesis, and a directed enhancement of adipocyte metabolism might have value in weight reduction. So it is important to know the different metabolic characteristics in human adults who have detected BAT. Therefore, the purpose of the investigators study is to compare different metabolic characteristics in the presence of brown adipose tissue in humans.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent 18FDG-PET/CT scan year between 2008-2010

Exclusion Criteria:

* History of cardiovascular disease (myocardial infarction, unstable angina, stroke, or cardiovascular revascularization)
* Diabetes
* Stage 2 hypertension
* Severe renal or hepatic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who underwent 18FDG-PET/CT scan year between 2008-2010.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2010-12; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
presence metabolic syndrome | 5 months

SECONDARY OUTCOMES:
BMI | 5 months
visceral fat area | 5 months
adipokines | 5 months
sarcopenia | 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- korea University Guro Hospital, Seoul, South Korea